CLINICAL TRIAL: NCT01994252
Title: Resynchronization/Defibrillation for Ambulatory Heart Failure Trial in Patients With Permanent Atrial Fibrillation
Acronym: RAFT-PermAF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RN00208414
Record Dates: First submitted 2013-11-08; First posted 2013-11-25 (Estimated); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Heart Disease; Congestive Heart Failure; Atrial Fibrillation
Keywords: defibrillator; cardiac resynchronization
MeSH Terms: conditions — Heart Diseases; Heart Failure; Atrial Fibrillation | interventions — Defibrillators, Implantable

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Optimal Medical therapy plus ICD (Active Comparator): Patients randomized to the (ICD) Implantable-Defibrillator-Cardioverter only group will receive an ICD + optimal medical therapy
  Interventions: Device: Optimal Medical therapy plus ICD
- Optimal Medical therapy plus CRT/ICD (Active Comparator): Patients randomized to the (ICD) Implantable-Defibrillator-Cardioverter plus cardiac resynchronisation therapy (CRT) group will receive an ICD + CRT and optimal medical therapy
  Interventions: Device: Optimal Medical therapy plus CRT/ICD

INTERVENTIONS:
Device: Optimal Medical therapy plus ICD
  Arms: Optimal Medical therapy plus ICD
Device: Optimal Medical therapy plus CRT/ICD
  Arms: Optimal Medical therapy plus CRT/ICD

SUMMARY:
Atrial fibrillation (AF) and heart failure (HF) are two common heart conditions that are encountered with an increase in death and suffering. When both these two conditions occur in a patient, the patient's prognosis is poor with a reduced quality of life and impaired heart function. These patients have enlarged hearts, specifically the left ventricle (major pumping chamber), which impairs the heart's pumping capacity, leading to symptoms such as fatigue, shortness of breath from any type of exertion, and swelling, usually of the feet and ankles.

In these HF patients who are in AF all of the time, who would otherwise be a suitable candidate for an implantable defibrillator to prevent sudden cardiac death, we would like to determine whether adding pacing of both ventricles will reduce heart size (left ventricular end systolic volume index LVESVi) as measured by ultrasound, which can improve its function and help the heart pump more efficiently.

Other studies have shown that adding pacing to both ventricles is of benefit in HF patients with mild to moderate symptoms and have a regular heart rhythm. The Investigators now want to explore if this therapy will benefit those patients with a permanent irregular heart rhythm (AF).

DETAILED DESCRIPTION:
Heart failure (HF) is increasing in prevalence and incidence and is the most common reason for hospital admissions of patients over the age of 65. Therapy for HF has evolved over the last two decades. Cardiac resynchronization therapy (CRT) is a therapy that attempts to resynchronize the sequence of ventricular contraction in heart failure (HF) patients with left ventricular (LV) systolic dysfunction and ventricular dyssynchrony. CRT is achieved by stimulating both RV and LV together, synchronized to right atrial excitation to achieve atrio-ventricular synchrony. Clinical trials have demonstrated that CRT reduced heart size, improved survival and reduced HF hospitalization in mild to advanced HF patients. This knowledge translated to a change in practice guidelines and the adoption of CRT into clinical practice benefitting many HF patients CRT is now an important state-of-the-art therapy for HF patients with LV systolic dysfunction, low LVEF, and prolonged QRS duration in sinus rhythm, since the vast majority of the CRT clinical research was performed in patients in sinus rhythm. However, in the ~25% of HF patients with permanent atrial fibrillation (AF), the effectiveness of CRT is not clear. It is therefore timely to address the question of whether the addition of CRT to optimal HF treatment, rate control and an ICD improves cardiac outcomes in individuals with heart failure (HF) and permanent atrial fibrillation (AF). The outcomes will be measured by a hierarchy of all-cause mortality, HF events, Left Ventricular Ejection Fraction (LVEF) and improvement in Quality of Life (QoL) in patients with permanent AF, mild to moderate HF, left ventricular (LV) systolic dysfunction, and prolonged QRS duration, when compared to implantable cardioverter defibrillator (ICD) therapy alone.

Objectives: To determine whether cardiac resynchronization therapy will improve cardiac outcomes for heart failure patients with permanent atrial fibrillation, mild to moderate heart failure, left ventricular systolic dysfunction, and prolonged QRS duration, when compared to implantable cardioverter defibrillator (ICD) therapy alone.

Methods: This is a multi-centre randomized controlled trial of two treatment groups. The patients, primary physicians and the heart failure caregivers will be blinded to the treatment allocation. The device follow-up caregivers will not be blinded. Patients with NYHA Class II and III HF symptoms, LVEF HF ≤ 35%, permanent AF, on optimal medical therapy and QRS durations ≥ 130 ms when the QRS morphology is LBBB, or QRS durations ≥ 150 ms when the QRS morphology is non-LBBB, or Paced QRS will be included in the trial. Patients should be suitable candidates for either of the 2 treatment strategies. There will be 200 patients randomized in 1:1 ratio to two groups: 1) ICD-CRT, 2) ICD only. All patients will undergo baseline clinical evaluation, echocardiogram measurements, quality of life assessment, medication assessment, and 6-minute walk distance.. The patients will be followed at 1 month, 3 months, 6 months and then every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NYHA Class II or III HF symptoms (assessment in the last 3 months)
* Permanent AF
* Optimal Medical Therapy for HF of at least 3 months (according to 2009 ACCF/AHA and ESC 2012 recommendations,)
* LVEF ≤ 35% (assessment in the last 6 months)
* Candidacy for an ICD for primary or secondary prevention of sudden cardiac death
* QRS durations ≥ 130 ms when the QRS morphology is LBBB, or QRS durations ≥ 150 ms when the QRS morphology is non-LBBB or Paced QRS

Exclusion Criteria:

* In-hospital patients who have acute cardiac or non-cardiac illness that requires intensive care
* Intra-venous inotropic agent in the last 4 days
* Patients with a life expectancy of less than one year from non-cardiac cause.
* Expected to undergo cardiac transplantation within one year (status I)
* Acute coronary syndrome (including MI) < 4 weeks
* Unable or unwilling to provide informed consent
* Uncorrected or uncorrectable primary valvular disease
* Restrictive, hypertrophic or reversible form of cardiomyopathy
* Severe primary pulmonary disease such as cor pulmonale
* Tricuspid prosthetic valve
* Patients included in other clinical trial that will affect the objectives of this study
* Coronary revascularization (CABG or PCI) < 3 months
* Patients with an existing ICD or CRT pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-08; Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is a hierarchy (winratio) of 1) all-cause mortality | 12 months
  Mortality data will be collected for the duration of the study
The primary outcome is a hierarchy (winratio) of 2) Heart Failure Events (>24 Hours admission for Heart Failure or clinically worsening Heart Failure leading to IV diuretics administered | 12 months
  HF events (> 24 hour admit or < 24 hr with IV diuretics) will be collected for the duration of the study
The primary outcome is a hierarchy (winratio) of 3) Left ventricular ejection fraction | baseline to 12 months
  Change in echocardiogram parameters LVEF measure
The primary outcome is a hierarchy (winratio) of 4) QoL - Minnesota Living with Heart Failure Questionnaire | baseline to 12 months
  Change in QoL MLHFQ. The MLHFQ score is used to measure quality of life. The MLHFQ consists of 21 questions answered on a 0-5 likert scale, with higher scores indicating a stronger impact of heart failure on QoL.

SECONDARY OUTCOMES:
All-cause mortality | Baseline to a minimum of 12 months
  Death all cause
Heart Failure Events | Baseline to a minimum of 12 months
  Admission to Hospital > 24 hrs for Heart Failure or <24 hrs with clinical worsending of HF leading to intervention
Changes in LVEF | Baseline to 12 months
  Left Ventricular ejection fraction
Quality of Life Questionnaire | Baseline to a minimum of 12 months
  Minnesota Living with Heart Failure
Composite of all-cause mortality and heart failure | Baseline to a minimum of 12 months
  All cause death and admission to to Hospital > 24 hours for Heart Failure
6 Minute walk distance | Baseline to a minimum of 12 months
  Hall walk distance over 6 minute timeframe
Cardiovascular mortality | Baseline to a minimum of 12 months
  Cardiovascular Death
Cost-effectiveness | Baseline to a minimum of 12 months
  Readmission for Heart Failure
Cardiovascular hospitalizations | Baseline to a minimum of 12 months
  Cardiovascular Admission to Hospital > 24 hours
Quality of Life Questionnaire | Baseline to a minimum of 12 months
  EQ5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Anthony SL Tang, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (15):
- Canada (15):
  - Libin Cardiovascular Institute of Alberta, Calgary, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Victoria Cardiac Arrhythmia Trials, Victoria, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Queen Elizabeth II Health Science, Halifax, Nova Scotia
  - Hamilton Health Sciences, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - St. Michael's General Hospital, Toronto, Ontario
  - CHUM Centre hospitalier universitaire de Montréal, Montreal, Quebec
  - McGill Health Science Centre, Montreal, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Quebec, Québec, Quebec
  - Le Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec

REFERENCES:
- [Background] Tang AS, Wells GA, Talajic M, Arnold MO, Sheldon R, Connolly S, Hohnloser SH, Nichol G, Birnie DH, Sapp JL, Yee R, Healey JS, Rouleau JL; Resynchronization-Defibrillation for Ambulatory Heart Failure Trial Investigators. Cardiac-resynchronization therapy for mild-to-moderate heart failure. N Engl J Med. 2010 Dec 16;363(25):2385-95. doi: 10.1056/NEJMoa1009540. Epub 2010 Nov 14. PMID 21073365